CLINICAL TRIAL: NCT05210543
Title: Acquisition and Long-term Observation of Patients With Severe Allergic Reactions
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Margitta Worm, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: Anaphylaxis Registry
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Anaphylaxis
MeSH Terms: conditions — Anaphylaxis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — option for Blood sampling (Serum, Blood cells, Cytokines, Biomarkers)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anaphylactic reaction (observational): Patients who experienced an anaphylactic reaction will be observed
  Interventions: Other: not applicable, observational study

INTERVENTIONS:
Other: not applicable, observational study — Patients do not receive intervention; observational study

SUMMARY:
The Anaphylaxis Registry aims to assess data in a standardized form about symptoms, triggers, cofactors and therapy management from patients who experienced an anaphylactic reaction. This should improve diagnosis and long-term management of these life-threatening allergic reactions.

DETAILED DESCRIPTION:
A better understanding of the triggers and pathology of anaphylactic reactions could lead to a better diagnosis and prophylaxis to avoid the occurence of these life-threatening allergic reactions. This can be an advantage for affected persons regarding the their treatment and long-term management.

The Anaphylaxis Registry is an opportunity to gather these standardized data. The blood sampling is optional for the patient, however, it will contribute to the better understanding of the sensitization profile and possible mechanisms. Recent publications showed a correlation between an anaphylactic reaction and certain biomarkers. Those data will be validated in a larger number of population with identification of further biomarkers. It is presumed that certain genetic and epigenetic polymorphisms are abundant for patients who experienced an anaphylaxis.

To summarize, this study aims to contribute to a better understanding of the anaphylaxis in general, the diagnosis, and the prognosis with different severities. With the identification of a certain trigger, the obtained understanding may help to decrease the risk of or prevent future repeating reactions.

ELIGIBILITY:
Inclusion Criteria:

* Anaphylactic reaction within the past 12 months

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who experienced a severe anaphylactic reaction and presenting in a participating center
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Influence of risk factors | 10 years
  Correlation between risk factors (age, epiphenomenon, comorbidity) and severity of anaphylaxis

SECONDARY OUTCOMES:
Epiphenomenon | 10 years
  Correlation between epiphenomenoa of the anaphylaxis and the frequency of allergic reactions
Current use of adrenaline | 10 years
  Assessment of acute treatments with adrenaline
Future use of adrenaline | 10 years
  Comparison of the frequencies of the use of adrenaline from beginning to end of the observation
Country-specific differences in anaphylaxis handling | 10 years
  Comparison of the triggers, diagnosis, treatment and prophylaxis of anaphylactic reactions throughout different countries
Biomarkers | 10 years
  Identification of biomarkers (e.g. PGE2 via ELISA, Tryptase via ImmunoCAP) for anaphylactic reactions
Epigenetics | 10 years
  Correlation of genetic and epigenetic factors with the pathogenesis of severe allergic reactions

CONTACTS AND LOCATIONS:
Overall Officials: Margitta Worm, Prof., Study Chair — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided